CLINICAL TRIAL: NCT04193540
Title: Evaluation of Decision Capacity of ICU Patients Under Sedatives. A Prospective Observational Multicenter Study.
Acronym: DexCap
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: DEXCAP
Record Dates: First submitted 2019-12-05; First posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Intensive Care Unit Patient; Mechanical Ventilation; Sedatives; Decision-making Capacity; Confusion
Keywords: Intensive Care Unit patient; Mechanical Ventilation; Sedatives; Decision-making capacity; Confusion
MeSH Terms: conditions — Confusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ACE questionnaire: Every patient under mechanical ventilation (intubated or tracheotomized), with or without sedatives, able to communicate and alert (RASS -1 to +1), and not delirious (CAM-ICU negative) will be assessed by Johns Hopkins ACE questionnaire by a person not in charge of the patient.
  Interventions: Other: ACE questionnaire

INTERVENTIONS:
Other: ACE questionnaire — Regardless of the result of the ACE questionnaire, physician, resident and nurse in charge of the patient will be asked their clinical opinion on decision-making capacity of the patient, based on a 4 steps Lickert scale and blindly of ACE result.

SUMMARY:
This prospective observational multicenter study is intended to investigate the impact of sedatives on the decision capacity of intensive care units patients.

DETAILED DESCRIPTION:
Medicine has recently turned from paternalism to patient-centered decisions giving them back autonomy to determine their own treatments and end-of-life directives. Main prerequisite is patient's competence to fully understand information given from medical staff, integrate it and resituate comprehensive willing.

Informed decision-making necessitates patient's ability to appropriately communicate and interact with its environment. Intensive care unit (ICU) patients are often intubated -rendering oral communication impossible- and get sedated with various medications (hypnotics and opioids). Despite an apparently appropriate communication, some of them are confused. Confusion is regularly under diagnosed in ICU settings and necessitates specific tools to be detected, such as CAM-ICU (Confusion Assessment Method in ICU). While not confused, a patient might lack decision-making capacity, meaning that despite obvious communication, more elaborated cognitive function remains uncertain and often inappropriate. Decision-making capacity can be evaluated with dedicated scores such as the Johns Hopkins adapted cognitive examination (ACE). This score has recently been formally translated into French.

The influence of sedatives on decision-making capacity remains unknown to date. This prospective observational multicentre study is intended to investigate the impact of sedatives on the decision-making capacity of ICU patients. Furthermore, each sub-score of the ACE (orientation, language, registration, attention and calculation, and recall) will be investigated according to sedatives types. Patients' decision-making capacity will be clinically assessed by physician, resident and nurse in charge, blindly of ACE result.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated patient (intubation or tracheotomy)
* Not delirious (negative CAM ICU)
* Calm and alert (RASS -1 to +1) since at least 12 hours and less than 72 hours
* Receiving sedatives and/or analgesics and/or medications interfering with neurological functions
* Adult patients with social security coverage

Exclusion Criteria:

* Brain injured patients (traumatic brain injury, ischemic or hemorrhagic stroke, sub-arachnoid hemorrhage, intra-parenchymal bleeding, hypoxic post cardiac arrest)
* Known cognitive disorders (MMSE < 20)
* Neurodegenerative disease
* Pregnant woman
* Protocol refusal by the patient or closest next-of-kin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every patient under mechanical ventilation (intubated or tracheotomized), with or without sedatives, able to communicate and alert (RASS -1 to +1), and not delirious (CAM-ICU negative) will be assessed by Johns Hopkins ACE questionnaire by a person not in charge of the patient.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-07-15 (Actual); Primary Completion 2020-07-15 (Estimated); Study Completion 2020-08-15 (Estimated)

PRIMARY OUTCOMES:
Decision-making capacity evaluated by Johns Hopkins ACE questionnaire | After inclusion
  Global decision-making capacity is evaluated by Johns Hopkins ACE with a 3 groups classification (< 29 severe alteration, 29-55: moderate alteration; > 55 light alteration or normal cognitive function).

SECONDARY OUTCOMES:
Decision-making capacity clinically evaluated by physician, resident and nurse in charge of the patient | : Immediately after inclusion and prior to Johns Hopkins ACE conduct
  Clinical determination of decision-making capacity of the patient blindly of Johns Hopkins ACE results
ACE sub-items | Immediately after inclusion
  Decision-making capacity sub-items as determined by ACE (orientation, language, registration, attention and calculation, and recall)
ICU length of stay | ICU discharge - Up to day 100
  ICU length of stay
Hospital length of stay | Hospital discharge - Up to day 200
  Hospital length of stay
Ventilatory free days | Hospital discharge - Up to day 200
  Ventilatory free days
Sedatives used within 72 hours before decision-making capacity evaluation | Within 72 hours before inclusion
  Sedatives administered to the patient within 72 hours before Johns Hopkins ACE will be collected (midazolam, propofol, dexmedetomidine, ketamine, halogenated volatile agents)
Analgesics used within 72 hours before decision-making capacity evaluation | Within 72 hours before inclusion
  Analgesics administered to the patient within 72 hours before Johns Hopkins ACE will be collected (morphine, remifentanil, sufentanyl, fentanyl)
Other molecules used within 72 hours before decision-making capacity evaluation | Within 72 hours before inclusion
  Other molecules administered to the patient within 72 hours before Johns Hopkins ACE will be collected (neuroleptics, benzodiazepines, hydroxyzine, clonidine, others)
Sedatives used during decision-making capacity evaluation | During inclusion
  Sedatives administered to the patient during Johns Hopkins ACE will be (midazolam, propofol, dexmedetomidine, ketamine, halogenated volatile agents)
Analgesics used during decision-making capacity evaluation | During inclusion
  Analgesics administered to the patient during Johns Hopkins ACE will be collected (morphine, remifentanil, sufentanyl, fentanyl
Other molecules used during decision-making capacity evaluation | During inclusion
  Other molecules administered to the patient during Johns Hopkins ACE will be collected (neuroleptics, benzodiazepines, hydroxyzine, clonidine, others

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Godet, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No